CLINICAL TRIAL: NCT01415076
Title: The Optimal Timing of Carbon Dioxide Insufflation During Colonoscopy in Unsedated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Peng-Jen Chen, Dr., Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TSGH-C99-062
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Outpatients
MeSH Terms: interventions — Insufflation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insertion without CO2 insufflation (Placebo Comparator): Patients were randomly allocated to receive whole procedure or extubation-only CO2 insufflation, using a randomized computer-generated list.
  Interventions: Procedure: Insufflation with CO2
- Insertion with CO2 (Experimental): Patients were randomly allocated to receive whole procedure or extubation-only CO2 insufflation, using a randomized computer-generated list.
  Interventions: Procedure: Insufflation with CO2

INTERVENTIONS:
Procedure: Insufflation with CO2 — Patients were randomly allocated to receive whole procedure or extubation-only CO2 insufflation, using a randomized computer-generated list.
  Other Names: the Olympus UCR Endoscopic CO2 Regulation Unit

SUMMARY:
Insufflation of carbon dioxide (CO2) instead of air can reduce pain resulting from colon distension after colonoscopy because CO2 is rapidly absorbed from the colon and excreted through the lungs. This reduces the effects of colonic distension and minimizes intracolonic gas at the end of the examination. The aims of the study were to evaluate the timing of administering CO2 insufflation and to identify predictors of discomfort for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients with an appropriate indication for colonoscopy were considered eligible.

Exclusion Criteria:

* Exclusion criteria included severe hematochezia, acute colonic pseudo-obstruction, known obstructive lesions, age <18 years, prior colon resection, fulminant colitis, chronic obstructive pulmonary disease requiring oxygen, and a medical history of CO2 retention. Patients that required only a partial colonoscopy or were unable to read or understand Chinese were also excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
abdominal pain during and after colonoscopy | One day
  Pain was recorded on a ten-point visual analog scale (0- no pain, 10- worst imaginable pain) at left-sided colonoscopic insertion, right-sided colonoscopic insertion, and at 1, 3, 6, and 24 hours postprocedure.

SECONDARY OUTCOMES:
delayed bleeding | One day
colonoscopic cecal intubation time | One day
completeness of intubation | One day
loop formation | One day

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Yuan Hsieh, MD.PhD, Study Chair — Division of Gastroenterology, Tri-Service General Hospital
Locations (1):
- Division of Gastroenterology, Tri-Service General Hospital, Taipei, Taiwan